CLINICAL TRIAL: NCT03108157
Title: Endometrial Scratch Effect on Pregnancy Rates When Performed During the Previous Cycle of Embryo Transfer in Patients Undergoing Egg-donation IVF
Brief Title: Endometrial Scratch Effect on Pregnancy Rates in Patients Undergoing Egg-donation IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procreatec (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, ALEXANDRA IZQUIERDO RODRIGUEZ, MD, Procreatec
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOSCRATCH
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Results first posted 2019-12-04 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: EMBRYO IMPLANTATION
Keywords: IVF; DONOR EGGS; ENDOMETRIAL SCRATCH; PIPELLE; ONGOING PREGNANCY

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: intervention group (Experimental): Patients will be performed an endometrial scratch with Pipelle Cournier 3 to 4 weeks before the embryo transfer and then they will follow the conventional preparation protocol to receive embryos coming from an egg donation treatment.
  Interventions: Procedure: Endometrial scratch
- GROUP B: no intervention group (No Intervention): Patients will receive the conventional preparation protocol to receive embryos coming from an egg donation treatment.

INTERVENTIONS:
Procedure: Endometrial scratch — Patients included in the study group will be performed an endometrial scratch with Pipelle Cournier 3 to 4 weeks before embryo transfer.
  Other Names: Scratching
  Arms: GROUP A: intervention group

SUMMARY:
Clinical trial about the effect of endometrial scratch on pregnancy rates in patients undergoing a treatment with in-vitro fertilization with donor eggs, when doing the endometrial biopsy during the cycle prior to the embryo transfer.

DETAILED DESCRIPTION:
The aim of this clinical trial is to investigate whether an endometrial scratch during the cycle prior to embryo transfer cycle is effective or not in increasing pregnancy rates. Previous studies about this issue have not shown clear conclusions about the effectiveness of this method.

The endometrial scratch is a simple technique that consists in performing a mild injury to all the internal walls of the uterus with a Pipelle Cournier.

To achieve the trial objective, all participating patients are randomly divided into two groups. Once patients decide to participate in the trial, they are assigned to each group according to the randomization list:

Group A: Patients with transfer of fresh embryos after taking an endometrium biopsy during the previous cycle and then following the conventional preparation protocol.

Group B: Patients with transfer of fresh embryos with the conventional preparation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female undergoing IVF treatment with donor eggs

Exclusion Criteria:

* Severe male factor ( less tan 2 million spermatozoa per ml )
* Uterine abnormalities

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Galindo, PhD, Study Director — Hospital Universitario 12 Octubre; Laura De la Fuente, PhD, Study Chair — Hospital Universitario 12 Octubre
Locations (1):
- Procreatec, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dain L, Ojha K, Bider D, Levron J, Zinchenko V, Walster S, Dirnfeld M. Effect of local endometrial injury on pregnancy outcomes in ovum donation cycles. Fertil Steril. 2014 Oct;102(4):1048-54. doi: 10.1016/j.fertnstert.2014.06.044. Epub 2014 Jul 23. PMID 25064410
- [Background] Potdar N, Gelbaya T, Nardo LG. Endometrial injury to overcome recurrent embryo implantation failure: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Dec;25(6):561-71. doi: 10.1016/j.rbmo.2012.08.005. Epub 2012 Sep 12. PMID 23063812
- [Background] Nastri CO, Lensen SF, Gibreel A, Raine-Fenning N, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2015 Mar 22;(3):CD009517. doi: 10.1002/14651858.CD009517.pub3. PMID 25803542
- [Background] Gibreel A, El-Adawi N, Elgindy E, Al-Inany H, Allakany N, Tournaye H. Endometrial scratching for women with previous IVF failure undergoing IVF treatment. Gynecol Endocrinol. 2015 Apr;31(4):313-6. doi: 10.3109/09513590.2014.994603. Epub 2015 Jan 5. PMID 25561347
- [Background] Ko JK, Ng EH. Scratching and IVF: any role? Curr Opin Obstet Gynecol. 2016 Jun;28(3):178-83. doi: 10.1097/GCO.0000000000000264. PMID 26950730
- [Background] Singh N, Toshyan V, Kumar S, Vanamail P, Madhu M. Does endometrial injury enhances implantation in recurrent in-vitro fertilization failures? A prospective randomized control study from tertiary care center. J Hum Reprod Sci. 2015 Oct-Dec;8(4):218-23. doi: 10.4103/0974-1208.170401. PMID 26752857
- [Background] Wise J. Endometrial scratching improves IVF pregnancy rate. BMJ. 2013 Oct 4;347:f6007. doi: 10.1136/bmj.f6007. No abstract available. PMID 24100512
- [Background] Yang R, Yang S, Li R, Chen X, Wang H, Ma C, Liu P, Qiao J. Biochemical pregnancy and spontaneous abortion in first IVF cycles are negative predictors for subsequent cycles: an over 10,000 cases cohort study. Arch Gynecol Obstet. 2015 Aug;292(2):453-8. doi: 10.1007/s00404-015-3639-8. Epub 2015 Feb 8. PMID 25663163
- [Background] Ueno J, Salgado RM, Tomioka RB, Colucci JA, Schor E, Carvalho FM. Clinical relevance of diagnostic hysteroscopy with concurrent endometrial biopsy in the accurate assessment of intrauterine alterations. Arch Gynecol Obstet. 2015 Aug;292(2):363-9. doi: 10.1007/s00404-015-3634-0. Epub 2015 Feb 3. PMID 25644507
- [Background] Timeva T, Shterev A, Kyurkchiev S. Recurrent implantation failure: the role of the endometrium. J Reprod Infertil. 2014 Oct;15(4):173-83. PMID 25473625
- [Background] Gnainsky Y, Granot I, Aldo P, Barash A, Or Y, Mor G, Dekel N. Biopsy-induced inflammatory conditions improve endometrial receptivity: the mechanism of action. Reproduction. 2015 Jan;149(1):75-85. doi: 10.1530/REP-14-0395. Epub 2014 Oct 27. PMID 25349438
- [Background] Lensen S, Martins W, Nastri C, Sadler L, Farquhar C. Pipelle for Pregnancy (PIP): study protocols for three randomised controlled trials. Trials. 2016 Apr 27;17(1):216. doi: 10.1186/s13063-016-1301-9. PMID 27121007
- [Background] Lensen S, Sadler L, Farquhar C. Endometrial scratching for subfertility: everyone's doing it. Hum Reprod. 2016 Jun;31(6):1241-4. doi: 10.1093/humrep/dew053. Epub 2016 Mar 22. PMID 27008891
- [Background] Karimzadeh MA, Ayazi Rozbahani M, Tabibnejad N. Endometrial local injury improves the pregnancy rate among recurrent implantation failure patients undergoing in vitro fertilisation/intra cytoplasmic sperm injection: a randomised clinical trial. Aust N Z J Obstet Gynaecol. 2009 Dec;49(6):677-80. doi: 10.1111/j.1479-828X.2009.01076.x. PMID 20070722
- [Background] Nastri CO, Polanski LT, Raine-Fenning N, Martins WP. Endometrial scratching for women with repeated implantation failure. Hum Reprod. 2014 Dec;29(12):2855-6. doi: 10.1093/humrep/deu257. Epub 2014 Oct 14. No abstract available. PMID 25316455
- [Background] Panagiotopoulou N, Karavolos S, Choudhary M. Endometrial injury prior to assisted reproductive techniques for recurrent implantation failure: a systematic literature review. Eur J Obstet Gynecol Reprod Biol. 2015 Oct;193:27-33. doi: 10.1016/j.ejogrb.2015.06.026. Epub 2015 Jul 17. PMID 26218557
- [Background] Kitaya K, Matsubayashi H, Takaya Y, Nishiyama R, Yamaguchi K, Ishikawa T. Clinical background affecting pregnancy outcome following local endometrial injury in infertile patients with repeated implantation failure. Gynecol Endocrinol. 2016 Jul;32(7):587-90. doi: 10.3109/09513590.2016.1144742. Epub 2016 Feb 18. PMID 26890618
- [Background] Nastri CO, Ferriani RA, Raine-Fenning N, Martins WP. Endometrial scratching performed in the non-transfer cycle and outcome of assisted reproduction: a randomized controlled trial. Ultrasound Obstet Gynecol. 2013 Oct;42(4):375-82. doi: 10.1002/uog.12539. Epub 2013 Sep 2. PMID 23754314
- [Derived] Izquierdo A, de la Fuente L, Spies K, Rayward J, Lopez L, Lora D, Galindo A. Endometrial scratch vs no intervention in egg donation cycles: the ENDOSCRATCH trial protocol. BMC Pregnancy Childbirth. 2020 May 30;20(1):333. doi: 10.1186/s12884-020-02958-0. PMID 32473654
- [Derived] Izquierdo Rodriguez A, de la Fuente Bitaine L, Spies K, Lora D, Galindo A. Endometrial Scratching Effect on Clinical Pregnancy Rates in Patients Undergoing Egg Donor In Vitro Fertilization Cycles: the ENDOSCRATCH Randomized Clinical Trial (NCT03108157). Reprod Sci. 2020 Oct;27(10):1863-1872. doi: 10.1007/s43032-020-00204-8. Epub 2020 May 28. PMID 32468267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on January 2017 and finished in October 2018. All patients were recruited at ProcreaTec Fertility Clinic in Madrid
Period: Overall Study
Arm/Group | GROUP A: Intervention Group | GROUP B: no Intervention Group
Started | 176 | 176
Completed | 161 | 172
Not Completed | 15 | 4
Not completed — Protocol Violation | 15 | 4

BASELINE CHARACTERISTICS:
Groups:
- GROUP B: Non Intervention Group: Patients will receive the conventional preparation protocol to receive embryos coming from an egg donation treatment.
- Total: Total of all reporting groups
Arm/Group | GROUP A: Intervention Group | GROUP B: Non Intervention Group | Total
Number analyzed (Participants) | 176 | 176 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.29 (4.27) | 41.50 (4.67) | 41.3 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 176 | 352
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 10 | 14
  White | 152 | 142 | 294
  More than one race | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 176 | 176 | 352
Smokers [Count of Participants; unit: Participants] | 34 | 29 | 63
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.78 (3.39) | 22.92 (3.31) | 22.8 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Positive Pregnancy Test
Description: Positive test (hcG>10 UI/ml)
Time Frame: 12 to 14 days after embryo transfer
Measure: Count of Participants; unit: Participants
Arm/Group | GROUP A: Intervention Group | GROUP B: no Intervention Group
Number analyzed (Participants) | 161 | 172
Participants | 112 | 113

2. Primary Outcome: Clinical Pregnancy
Description: Ultrasound confirmation of intrauterine pregnancy
Time Frame: 5 weeks of pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | GROUP A: Intervention Group | GROUP B: no Intervention Group
Number analyzed (Participants) | 161 | 172
Participants | 104 | 102

3. Secondary Outcome: Live Birth
Description: Birth after 24 weeks of pregnancy
Time Frame: Pregnancy beyond 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GROUP A: Intervention Group | GROUP B: no Intervention Group
Number analyzed (Participants) | 161 | 172
Participants | 92 | 85

ADVERSE EVENTS:
Time Frame: Adverse effects will be controlled for every patient for 12 months, starting on the day of randomization.
Description: All-Cause Mortality and Serious and Non-serious Adverse Events were monitored since all patients were followed up and contacted to assess the results of their pregnancies and determine the possible negative events. In our population no deaths or Serious Adverse Events were observed.
  We did not observe any Mortality or Adverse Events related to the intervention, since this intervention does not differ from conventional clinical practice.
Arm/Group | GROUP A: Intervention Group | GROUP B: no Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/172
Other Adverse Events (participants affected / at risk) | 36/161 | 47/172
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GROUP A: Intervention Group (N=161) | GROUP B: no Intervention Group (N=172)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 12 | 12 — Pregnancy loss before 12th week of gestation.
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 3 — Extrauterine evidence of pregnancy
Vanishing twin (Pregnancy, puerperium and perinatal conditions) | 3 | 3 — Second twin arrest before week 12th of gestation
Placentation abnormalities (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Alterations in placental development (accretism, percretism...)
Intrauterine growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Pathological decrease in the growth of the fetus
Preterm delivery threat (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Menace of preterm before the 37th week of gestation
Premature membrane rupture (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Rupture of gestational membranes before the 37th week of pregnancy.
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 2 | 1 — Presence of a diabetical status in a pregnant woman who was not previously diabetic
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 4 | 6 — Gestational hypertension and proteinuria
Gestational cholestasis (Pregnancy, puerperium and perinatal conditions) | 1 | 1 — Biliary acid alteration due to gestational status
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Voluntary interruption of gestation
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 12 | 16 — Delivery before the 37th week of pregnancy
2nd twin stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 2 — Intrauterine death of the 2nd twin before delivery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03108157/SAP_001.pdf
  • Study Protocol (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT03108157/Prot_002.pdf